CLINICAL TRIAL: NCT01603992
Title: Quitting Marijuana Use: Self-Report Study of Quitting Strategies and Withdrawal Symptoms
Brief Title: Quiting Marijuana Use: Self-report Study of Quitting Straegies and Withdrawal Symptoms
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906408; 06-DA-N408; NCT00679016 (obsolete NCT alias)
Record Dates: First submitted 2012-05-19; First posted 2012-05-23 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2012-05-03

CONDITIONS: Cannabis Abuse; Cannabis Dependence
Keywords: Cannabis; Craving; Questionnaire; Non-Treatment; Drug Use
MeSH Terms: conditions — Marijuana Abuse

SUMMARY:
Background:

- Marijuana is the most widely used illicit drug in the world, yet relatively little is known about users who try to quit without formal treatment ( spontaneous quitting). Studies have suggested that there are some common strategies that many individuals use in spontaneous quitting, such as changing one s lifestyle or identity, reminding oneself of negative consequences, support from family and friends, and religion. However, more research is needed to determine potential treatment strategies for marijuana use.

Objectives:

* To identify strategies used to help with marijuana quitting among non-treatment seeking adult marijuana users.
* To identify withdrawal symptoms experienced during marijuana quitting and their relationship to the quitting strategies used and the outcome of the quit attempt.
* To evaluate whether subgroups of marijuana users differ in their experience of marijuana quitting.

Eligibility:

- Individuals at least 18 years of age who have made at least one attempt to quit marijuana use.

Design:

* The study will consist of one visit of approximately 1 to 2 hours.
* Participants will fill out three questionnaires. The questionnaires have different types of questions, and will ask about background and lifestyle, marijuana use and craving patterns and behaviors, and difficulties in previous attempts to quit using marijuana.

DETAILED DESCRIPTION:
Marijuana is the most widely used illicit drug in the world, yet relatively little is known about users who try to quit without formal treatment (so-called spontaneous quitting). This study will use two self-report questionnaires to collect information on the socio-demographic characteristics, marijuana use history, most difficult marijuana quit experience, and marijuana craving from a convenience sample of 1230 adult, non-treatment-seeking marijuana users. The questionnaires take 45-60 minutes to administer. Data will be analyzed for patterns and correlations among the characteristics of the quit attempt, including any withdrawal symptoms, quitting strategies used, and its success. The marijuana craving data will be analyzed to evaluate the validity of this measure of marijuana craving. There are no direct benefits to subjects from study participation. The scientific benefit is an improved understanding of spontaneous quitting of marijuana use, which may lead to improved interventions for marijuana users in the future. There are no physical risks to subjects. There are risks of anxiety or embarrassment while taking the questionnaire and of loss of confidentiality of sensitive information collected about subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. age 18 or older
  2. have made at least one attempt to quit marijuana use
  3. able to give valid informed consent
  4. ability to understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 822 (Actual)
Dates: Start 2005-11-08; Study Completion 2012-05-03

PRIMARY OUTCOMES:
Marijuana Quit Questionnaire | 1 to 2 hours

SECONDARY OUTCOMES:
Marijuana Craving Questionnaire, and Additional Questions about Marijuana Craving

CONTACTS AND LOCATIONS:
Overall Officials: David A Gorelick, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (3):
- United States (3):
  - National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland
  - Maryland Psychiatric Research Center (MPRC) 55 Wade Avenue, Catonsville, Maryland
  - Medical University of S. Carolina, Charleston, South Carolina

REFERENCES:
- [Background] Adamson SJ, Sellman JD. A prototype screening instrument for cannabis use disorder: the Cannabis Use Disorders Identification Test (CUDIT) in an alcohol-dependent clinical sample. Drug Alcohol Rev. 2003 Sep;22(3):309-15. doi: 10.1080/0959523031000154454. PMID 15385225
- [Background] Boyd SJ, Tashkin DP, Huestis MA, Heishman SJ, Dermand JC, Simmons MS, Gorelick DA. Strategies for quitting among non-treatment-seeking marijuana smokers. Am J Addict. 2005 Jan-Feb;14(1):35-42. doi: 10.1080/10550490590899835. PMID 15804875
- [Background] Budney AJ, Hughes JR, Moore BA, Vandrey R. Review of the validity and significance of cannabis withdrawal syndrome. Am J Psychiatry. 2004 Nov;161(11):1967-77. doi: 10.1176/appi.ajp.161.11.1967. PMID 15514394
- [Derived] Koola MM, Boggs DL, Kelly DL, Liu F, Linthicum JA, Turner HE, McMahon RP, Gorelick DA. Relief of cannabis withdrawal symptoms and cannabis quitting strategies in people with schizophrenia. Psychiatry Res. 2013 Oct 30;209(3):273-8. doi: 10.1016/j.psychres.2013.07.044. Epub 2013 Aug 20. PMID 23969281
- [Derived] Boggs DL, Kelly DL, Liu F, Linthicum JA, Turner H, Schroeder JR, McMahon RP, Gorelick DA. Cannabis withdrawal in chronic cannabis users with schizophrenia. J Psychiatr Res. 2013 Feb;47(2):240-5. doi: 10.1016/j.jpsychires.2012.10.010. Epub 2012 Nov 10. PMID 23146560